CLINICAL TRIAL: NCT02886806
Title: Fully Automated Anesthesia, Analgesia and Fluid Management Using Multiple Physiologic Closed-Loop Systems in High-Risk Vascular Surgery: a Pilot Study
Brief Title: Fully Automated Anesthesia, Analgesia and Fluid Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Hopital Foch (Other)
Responsible Party: Principal Investigator, Luc Barvais, Professor and head of the cardiothoracic and vascular anesthesia Clinics, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2016/328
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: General Anesthetic Drug Overdose; Adverse Effect of Intravenous Anesthetics, Sequela; Complication of Anesthesia; Drug Delivery System Malfunction; Hemodynamic Instability; Underdosing of Other General Anesthetics
Keywords: closed loop; remifentanil; propofol
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high risk vascular surgery (Experimental): Patients scheduled for high risk vascular surgery under automated total closed loop intravenous anesthesia and fluid management
  Interventions: Other: BIS XP, Covidien, Ireland; Other: EV-1000 TM, Edwards Lifesciences, Irvine, California, USA

INTERVENTIONS:
Other: BIS XP, Covidien, Ireland — Closed loop for propofol and remifentanil using BIS XP TM, Covidien, Ireland
  Other Names: bispectral index
Other: EV-1000 TM, Edwards Lifesciences, Irvine, California, USA — Closed loop for fluid perfusion using EV-1000 TM, Edwards Lifesciences, Irvine, CA, USA

SUMMARY:
Evaluate the feasibility and quality of automated anesthesia, analgesia and fluid management based on a combination of several physiological variables (bispectral index [BIS], stroke volume [SV], and stroke volume variation [SVV]) using 2 independent physiologic closed-loop systems (PCLS) in patients undergoing high risk vascular surgery

DETAILED DESCRIPTION:
Evaluate the feasibility and quality of automated anesthesia, analgesia and fluid management based on a combination of several physiological variables (bispectral index [BIS], stroke volume [SV], and stroke volume variation [SVV]) using 2 independent physiologic closed-loop systems (PCLS) in patients undergoing high risk vascular surgery.

All patients will receive total intravenous anesthesia in target controlled infusion mode using the population pharmacokinetic sets of Schnider for propofol and Minto for remifentanil to target the effect-site concentration. Infusion Toolbox 95 version 4.11 software (Free University of Brussels, Brussels, Belgium) implemented in a personal computer serving as a platform for: calculating effect-site concentrations of propofol and remifentanil; displaying effect-site concentration estimates in real time; providing a user interface that permits entry of patients' demographic data (sex, age, weight, and height) and modifications to target concentrations; controlling the propofol and remifentanil infusion pumps (Alaris Medical, Hampshire, United Kingdom); and recording calculated effect-site drug concentrations.

All patients will receive a baseline crystalloid infusion (PlasmaLyte, Baxter, Belgium) delivered by a pump at a rate of 3 mL/ kg/h (Fresenius Kabi, Belgium). Additional fluid was given using a goal-directed fluid therapy protocol guided by the cardiac output monitor (EV-1000; Edwards Lifesciences) and consisted of 100 mL boluses (Voluven, Fresenius Kabi, Germany) delivered by our PCLS (Learning Intravenous Resuscitator [LIR]). For fluid output, a Q-Core Sapphire Multi-Therapy Infusion Pump (Q-Core, Israel) was controlled by the LIR using software provided by Q-Core via a serial connection (Commands Server R.01). If hypotension occurred (defined as mean arterial pressure <20% of baseline blood pressure) and no fluid is delivered by the LIR, it will be treated by the anesthesiologist using a vasopressor drug.

In this pilot study, each closed loop also will operate independently, guided only by its own respective inputs (BIS for the propofol; SV and SVV for the fluid boluses).

The investigators will also measure analgesia using the PhysioDoloris monitoring device (MDoloris Medical Systems, Lille, France).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for high risk vascular surgery
* Patients American Society Anesthesiologist classification: 3 or 4

Exclusion Criteria:

* age less than 18 years,
* patients with arrhythmias like atrial fibrillation
* allergy to latex, propofol, remifentanil, morphine, muscle relaxant or any of the excipients,
* pregnant woman
* combined general and regional anesthesia,

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The percentage of adequate anesthesia defined as a BIS between between 40 and 60, a SVV < 13% and/or cardiac index > 2.5 litre/min/m² for more/equal of 85% of the surgical time | at time of surgery

SECONDARY OUTCOMES:
Drug consumption: remifentanil dose | at time of surgery
Drug consumption: propofol dose | at time of surgery
amount of fluid given | at time of surgery
number of automatic modifications of the propofol and remifentanil concentrations | at time of surgery
number of patients movements | at time of surgery
number of hemodynamic abnormalities requiring treatment | at time of surgery
time to tracheal extubation | at time of surgery
intraoperative awareness | postoperative day 1 or 2
Occurrence of burst suppression | at time of surgery
Need for anesthetist interventions over the system during the surgery | at time of surgery
performance of the closed-loop system | at time of surgery
Interactions between both closed-loop system during the intraoperative period especially during hypotension episodes | at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Luc Barvais, MD PhD, Study Director — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided